CLINICAL TRIAL: NCT01040273
Title: Management of Postoperative Pain After Total Hip Arthroplasty
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THA
Record Dates: First submitted 2009-12-20; First posted 2009-12-29 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Experiment (Experimental): Anesthetics intraarticular injection
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): saline intraarticular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacaine
  Arms: Experiment
Drug: Placebo
  Arms: Placebo

SUMMARY:
Orthopedic surgery is reportedly among the most painful surgical procedures. Surgical damage following major orthopedic surgery often involves a large, deep incision with considerable tissue dissection and muscle, bone, and vascular exposure. Post-operative pain after such surgery is exacerbated on movement or by reflex spasms of the muscles, which may delay mobilization, reduce satisfaction, prolong hospitalization, and possibly increase medical costs.

We design a prospective randomized study for postoperative pain control following total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for surgery of osteoarthritis of hip
* ability to tolerate surgery under general anesthesia.

Exclusion Criteria:

* refusal or the lack of mental ability to provide informed consent
* neuropathic pain or sensory disorders in the leg requiring surgery
* previous surgery of the hip joint
* coagulation abnormalities
* severe renal or hepatic impairment
* chronic opioid users
* known history of intolerance to the drugs used in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pain VAS score | pre-operaton, immediately post operation, postop 6hrs, postop 12hrs, postop 18hrs, postop 24hrs, post op 48hrs, postop 72hrs

SECONDARY OUTCOMES:
Functional score: WOMAC hip score, SF-36 | Pre-operation, immediately post-operation, postop 6 weeks, postop 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kweishian, Taoyuan, Taiwan

REFERENCES:
- [Derived] Chen DW, Hu CC, Chang YH, Lee MS, Chang CJ, Hsieh PH. Intra-articular bupivacaine reduces postoperative pain and meperidine use after total hip arthroplasty: a randomized, double-blind study. J Arthroplasty. 2014 Dec;29(12):2457-61. doi: 10.1016/j.arth.2013.12.021. Epub 2013 Dec 19. PMID 24439998